CLINICAL TRIAL: NCT00278369
Title: A Pilot Study of Denileukin Diftitox in Combination With High-Dose IL-2 for Patients With Metastatic Renal Cell Carcinoma
Brief Title: Pilot Study of Denileukin Diftitox Plus High-Dose IL-2 for Patients With Metastatic Renal Cancer
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: Northwestern University (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, Timothy Kuzel, Timothy Kuzel, MD, Northwestern University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NU 04U1; P30CA060553 (NIH); NU-04U1; STU00006770 (Other: Northwestern University IRB)
Record Dates: First submitted 2006-01-16; First posted 2006-01-18 (Estimated); Last update posted 2013-05-22 (Estimated); Status verified 2013-05

CONDITIONS: Kidney Cancer
Keywords: recurrent renal cell cancer; stage IV renal cell cancer; clear cell renal cell carcinoma
MeSH Terms: conditions — Kidney Neoplasms; Carcinoma, Renal Cell | interventions — aldesleukin; Interleukin-2; denileukin diftitox

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- A (Experimental): 6 mcg/kg Denileukin Diftitox administered IV/daily on days 8-10 of standard interleukin 2 dose course
  Interventions: Biological: aldesleukin; Biological: denileukin diftitox
- B (Experimental): 9 mcg/kg Denileukin Diftitox administered IV/daily on days -4 to -2 of standard interleukin 2 dose course
  Interventions: Biological: aldesleukin; Biological: denileukin diftitox
- C (Experimental): 9 mcg/kg Denileukin Diftitox administered IV/daily on days 8-10 of standard interleukin 2 dose course
  Interventions: Biological: aldesleukin; Biological: denileukin diftitox

INTERVENTIONS:
Biological: aldesleukin — The IL-2 is given as a 15-minute infusion through an intravenous catheter (I.V.), a small plastic tube that is put into your vein for the time you are receiving the study treatment. IL-2 is given through the I.V. once every 8 hours for 5 days (days 1-5). A second 5 day cycle of IL-2 will begin on the 15th day (days 15-19). This is one complete cycle (days 1-19) of IL-2 treatment
  Other Names: IL-2; Interleukin-2; Proleukin
Biological: denileukin diftitox — Denileukin diftitox will be administered once daily as a 15 to 60 minute infusion for 3 consecutive days.
  Other Names: ONTAK (denileukin diftitox); DAB 389 IL-2

SUMMARY:
RATIONALE: Combinations of biological substances in denileukin diftitox may be able to carry tumor-killing substances directly to kidney cancer cells. Interleukin-2 may stimulate the white blood cells to kill kidney cancer cells. Giving denileukin diftitox together with interleukin-2 may kill more tumor cells.

PURPOSE: This randomized phase I trial is studying the side effects of denileukin diftitox and interleukin-2 in treating patients with metastatic kidney cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* Determine the toxic effects of denileukin diftitox and high-dose interleukin-2 in patients with metastatic renal cell cancer.

Secondary

* Perform transforming growth factor (TGF)-beta promoter and TGF-beta receptor genotyping to search for variants that may be associated with tumor response to therapy.
* Determine the overall response rate (partial and complete) in patients treated with this regimen.
* Determine the time to progression in patients treated with this regimen.

OUTLINE: This is a randomized, pilot study.

The first 3 patients enrolled in the study receive high-dose interleukin-2 (IL-2) IV over 15 minutes, 3 times daily, on days 1-5 and 15-19 and denileukin diftitox IV over 15-60 minutes once daily on days 8-10. If no dose-limiting toxicity occurs after receiving denileukin diftitox, subsequent patients are randomized to 1 of 2 treatment arms.

* Arm I: Patients receive denileukin diftitox (at a higher dose than for the first 3 patients enrolled in the study) IV over 15-60 minutes once daily on days -4 to -2 and high-dose IL-2 IV over 15 minutes, 3 times daily, on days 1-5 and 15-19.
* Arm II: Patients receive high-dose IL-2 as in arm I and denileukin diftitox (at a higher dose than for the first 3 patients enrolled in the study) IV over 15-60 minutes at a higher dose once daily on days 8-10.

All patients may receive additional treatment with IL-2 alone in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed periodically for at least 4 years.

PROJECTED ACCRUAL: A total of 13 patients will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Documented histologically confirmed metastatic renal cell carcinoma

  * Clear cell histology
* Disease must be measurable as defined by lesions that can be accurately measured in at least one dimension with longest diameter > 20 mm using conventional techniques or > 10 mm with spiral CT scan

  * Must have at least one measurable lesion
  * If the measurable disease is restricted to a solitary lesion, its neoplastic nature should be confirmed by cytology/histology
  * Clinical lesions will only be considered measurable when they are superficial (e.g., skin nodules and palpable lymph nodes)
  * The following are considered nonmeasurable lesions:

    * Bone lesions
    * Leptomeningeal disease
    * Ascites
    * Pleural/pericardial effusion
    * Inflammatory breast disease
    * Lymphangitis cutis/pulmonis
    * Cystic lesions
    * Abdominal masses not confirmed and followed by imaging techniques
* No CNS metastases

PATIENT CHARACTERISTICS:

* ECOG performance status < 2
* Life expectancy of at least 4 months
* Serum creatinine < 2.0 mg/dL OR creatinine clearance > 50 mL/min
* Total bilirubin normal
* Platelets > 100,000/mm³
* WBC > 3,500/mm³
* No evidence of congestive heart failure
* No symptoms of coronary artery disease
* No serious cardiac arrhythmias
* A pretreatment cardiac stress test must be performed within 42 days of IL-2 treatment if any cardiac symptoms are present (patients with documented ischemia on the pretreatment cardiac stress test will be excluded from the study)
* Adequate pulmonary reserve

  * Pulmonary function tests (PFTs) must be performed within 42 days of IL-2 treatment

    * FEV_1 > 2.0 liters of > 75% predicted for height and age
    * Patients unable to perform PFTs will be excluded
* Women who are pregnant or lactating are not eligible
* Women of childbearing potential and sexually active males must commit to the use of effective contraception while on study
* Negative pregnancy test
* No known HIV-positive patients
* No evidence of active infection requiring antibiotic therapy
* Must not have a contraindication to treatment with pressor agents
* Must not have any significant medical disease that, in the opinion of the investigator, may interfere with completion of the study
* No history of another malignancy within the past 5 years other than basal cell skin cancer

PRIOR CONCURRENT THERAPY:

* Recovered from all toxic effects of prior therapy
* Must not currently receive chronic medication for asthma
* No prior interleukin-2 (IL-2) therapy
* No prior organ allografts
* No systemic corticosteroids in the 4 weeks prior to treatment
* No concurrent systemic steroids
* No radiotherapy, chemotherapy, or immunotherapy in the 4 weeks prior to the first dose of study treatment
* No concurrent radiotherapy, chemotherapy, or other immunotherapy
* No previous investigational agent within 4 weeks prior to the start of study treatment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2005-04; Primary Completion 2009-06 (Actual); Study Completion 2010-09 (Actual)

PRIMARY OUTCOMES:
The primary objective is to assess for toxicity | After each cycle of therapy and 30 days after the last treatment.
  To assess the toxicity

SECONDARY OUTCOMES:
The secondary objectives are to investigate differences in peak and duration of the expansion of CD4+, CD8+, CD4+CD 25+ and CD56+(dim and bright)CD25+ cells | Follow-up measurements must have met the SD criteria at least once after study entry at a minimum interval of 8 weeks.
  To investigate differences in peak and duration.
To investigate the effects of denileukin diftitox in combination with IL-2 on plasma TGF-beta levels | Cohort 1: Denileukin diftitox dose of 6μg/kg/ Days 1, 2, 3, 4, and 5. Cohort 2 Denileukin diftitox dose of 9μg/kg given 4, 3, 2, and 1 days prior to 1st day of each cycle. Cohort 3: Denileukin diftitox dose of 9μg/kg given days 8 and 9.
  To investigate the effects of denileukin diftitox
To perform TGF-beta promoter and TGF-beta receptor genotyping prior to the start of treatment to search for variants that may be associated with tumor response to therapy. | Cohort 1: Plasma TGF-beta levels to be given on day. Cohort 2: plasma TGF-beta levels to be given at day 1. Cohort 3: plasma TGF-beta levels given on days 1 through 5.
  To perform TGF-beta promoter and TGF-beta receptor genotyping
Overall response rate and time to progression | CT scans and other pertinent studies will be performed at week 10 to assess response.
  Overall response rate will be assessed.

CONTACTS AND LOCATIONS:
Overall Officials: Timothy M. Kuzel, MD, Study Chair — Robert H. Lurie Cancer Center
Locations (1):
- Robert H. Lurie Comprehensive Cancer Center at Northwestern University, Chicago, Illinois, United States